CLINICAL TRIAL: NCT00802711
Title: Phase II Randomised Clinical Trial of Accelerated Partial Breast Irradiation (APBI) Comparing 3-Dimensional Conformal Radiation Therapy and Multi-Catheter Interstitial Brachytherapy.
Brief Title: 3-Dimensional Conformal Radiation Therapy or Internal Radiation Therapy After Breast-Conserving Surgery in Treating Women With Stage I or Stage II Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-33 ICORG; ICORG-06-33; EU-20888
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; invasive ductal breast carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast | interventions — Radiotherapy, Conformal; Brachytherapy

ARMS (2):
- Arm I (Experimental): Patients undergo accelerated partial breast irradiation (APBI) using 3-dimensional conformal radiation therapy twice daily over 5-10 days (total of 10 fractions) in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-dimensional conformal radiation therapy
- Arm II (Experimental): Patients undergo APBI using multi-catheter interstitial brachytherapy twice daily over 5-10 days (total of 10 fractions) in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: brachytherapy

INTERVENTIONS:
Radiation: 3-dimensional conformal radiation therapy — Given twice a day for 10 fractions
  Arms: Arm I
Radiation: brachytherapy — Given twice a day for 10 fractions
  Arms: Arm II

SUMMARY:
RATIONALE: Specialized radiation therapy, such as 3-dimensional conformal radiation therapy, that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. Giving these treatments after surgery may kill any tumor cells that remain after surgery. It is not yet known whether 3-dimensional conformal radiation therapy is more effective than internal radiation therapy when given after surgery in treating early-stage breast cancer.

PURPOSE: This randomized phase II trial is studying 3-dimensional conformal radiation therapy to see how well it works compared with internal radiation therapy when given after breast-conserving surgery in treating women with stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the rate of successfully delivered accelerated partial breast irradiation (APBI) using 3-dimensional conformal radiation therapy vs multi-catheter interstitial brachytherapy in women with stage I or II invasive ductal carcinoma of the breast.
* To establish potential patient participation in ongoing phase III clinical trials (e.g., NSABP-B-39, GEC-ESTRO, RAPID, MPORT, and IRMA) that compare APBI to standard whole-breast irradiation.

Secondary

* To assess acute radiation-induced toxicity in these patients as assessed by NCI CTCAE version 3.0.
* To assess long-term radiation-induced toxicity in these patients as assessed by RTOG-EORTC scale.
* To assess the incidence and type of adverse events in the breast of these patients.
* To assess the incidence and type of procedure-related complications in these patients.
* To determine local control and pattern of recurrence in these patients.
* To determine disease-free survival (distant and recurrence-free survival) of these patients.
* To determine overall survival of these patients.
* To assess cosmesis in these patients as assessed by the Breast Cancer Treatment Outcome and RTOG scales.
* To assess treatment-related symptoms in these patients as assessed by the Breast Cancer Treatment Outcome scale.

OUTLINE: Patients are randomized to 1 of 2 treatment arms. Patients with a lumpectomy cavity/whole breast ratio 25-30% are assigned to treatment in arm II.

* Arm I: Patients undergo accelerated partial breast irradiation (APBI) using 3-dimensional conformal radiation therapy twice daily over 5-10 days (total of 10 fractions) in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo APBI using multi-catheter interstitial brachytherapy twice daily over 5-10 days (total of 10 fractions) in the absence of disease progression or unacceptable toxicity.

Patients complete quality-of-life questionnaires at baseline, on the last day of treatment, at 4 and 24 weeks after completion of treatment, and then annually for 3 years.

After completion of study treatment, patients are followed periodically for at least 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically proven invasive ductal carcinoma of the breast

  * Stage I or II disease (pathological tumor size ≤ 3 cm, N0, M0 disease)

    * No T2 (tumor size > 3 cm) or T3 disease
    * No lymph node (L0) or hemangiosis (V0) invasion
* Unilateral, unifocal, and unicentric tumor without associated suspicious diffuse microcalcification in the ipsilateral or contralateral breast

  * No multifocal/multicentric disease
* Previously treated with breast-conserving surgery with adequate axillary node management

  * Negative surgical resection margins for tumor (invasive tumor or ductal carcinoma in situ [DCIS]) on histology
  * Clearly identified primary tumor excision cavity (clips recommended) with a target lumpectomy cavity/whole breast ratio quantifiable and ≤ 25% on the post-operative CT scan

    * Patients with a lumpectomy cavity/whole breast ratio 25-30% are eligible but will undergo partial breast irradiation using multi-catheter interstitial brachytherapy during study
* Breast size amenable to partial breast irradiation (i.e., > A-cup size)
* No other pathological invasive tumor or DCIS
* No associated extensive DCIS component (< 25%)
* No associated Paget's disease of the nipple
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No breast implants
* No collagen vascular disease
* No psychiatric condition or other condition that, in the opinion of the investigator, would preclude study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy
* No concurrent chemotherapy

  * Sequential chemotherapy allowed
* Concurrent hormonal therapy allowed

Ages: 50 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Rate of successfully delivered accelerated partial breast irradiation | Never established as trial terminated

SECONDARY OUTCOMES:
Local control and pattern of recurrence | Never established as trial terminated
Disease-free survival (distant and recurrence-free survival) | Never established as trial terminated
Overall survival | Never established as trial terminated
Quality of life (e.g., cosmesis and treatment-related symptoms) as assessed by the Breast Cancer Treatment Outcome and RTOG scales | Never established as trial terminated
Acute radiation-induced toxicity as assessed by NCI CTCAE v3.0 | Never established as trial terminated
Long-term radiation-induced toxicity as assessed by RTOG-EORTC scale | Never established as trial terminated
Incidence and type of adverse events in the breast | Never established as trial terminated
Incidence and type of procedure-related complications | Never established as trial terminated

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Thirion, MD, Principal Investigator — Saint Luke's Hospital
Locations (1):
- Saint Luke's Radiation Oncology Network, Dublin, Ireland